CLINICAL TRIAL: NCT06110039
Title: Comparative Effects of Cervicothoracic Junction Mobilization With Arm Movements and Upper Thoracic Manipulation in Patients With Subachromial Impinegment Syndrome
Brief Title: Comparative Effects of Cervicothoracic Junction Mobilization and Thoracic Manipulation in Subachromial Impinegment Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S22C14G30039
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Subacromial Impingement Syndrome
Keywords: shoulder pain; NECK PAIN; UPPER THORACIC MOBILIZATION; CERVICOTHORACIC MOBILIZATION; SUBACROMIAL IMPIGEMENT SYNDROME
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Cervicothoracic junction mobilization with arm movement along with baseline treatment (Experimental)
  Interventions: Other: Cervicothoracic Junction Mobilization
- Group 2: upper thoracic manipulation woth baseline treatment (Experimental)
  Interventions: Other: Upper Thoracic Spine Manipulation:

INTERVENTIONS:
Other: Cervicothoracic Junction Mobilization — The therapist stood in back of the subject, who was seated straight on a chair. The therapist positioned the medial side of one hand's thumb. The desired level of vertebra can be strengthened by placing the index finger of the opposite hand on the spinous process. A pure transverse glide was executed from the affected side to the unaffected side.
  Arms: Group 1: Cervicothoracic junction mobilization with arm movement along with baseline treatment
Other: Upper Thoracic Spine Manipulation: — The therapist placed one hand on the patient's head and the hypothenar or thenar eminence of the other hand was placed over the T1 transverse process (the therapist's left hand was used for thrusting and vice versa for treating the left T1 Transverse process). As the tissue deficiency is taken up localizing the forces, the patient was urged to breathe in and out multiple times. While holding the hand on the head steady, a minor relative rotation in the opposite direction was caused, which led to the introduction of the postero-anterior force on the transverse process of T1(29). Patients will receive three sessions a week on alternate days for three weeks and follow up data will be taken once after completion of all three sessions using data collection tools
  Arms: Group 2: upper thoracic manipulation woth baseline treatment

SUMMARY:
The aim of this study is to investigate the comparative effects of high velocity low amplitude thrust manipulation of upper thoracic spine and spinal mobilization with arm movement on the subjects with the subacromial impingement syndrome.

DETAILED DESCRIPTION:
Subacromial impingement is the condition, in which the tissue underlying subacromial spaces are compressed between the head of the humerus and the acromion, is one ofthe main diagnoses of shoulder pain. Subjects frequently experience pain when engaging in anyoverhead activity.In general, medical practice, pain in the glenohumeral region is commonmusculoskeletal problem has almost 48% prevalence. Cervicothoracic junction refers to atherapeutic technique or manual therapy approaches that focuses on improving mobility andfunction in this area where the cervical neck and upper back spine meet. Upper thoracic manipulation refers to a manual technique used to address dysfunctions or restrictions in the upper portion of the thoracic vertebral region, which is the area of the thoracic vertebrae located between the cervical and mid back regions.Previously, studies were conducted individually to determine effectiveness of upper thoracic mobilization and cervico-thoracic mobilization with arm movement for treatment of subacromial bursitis. However, fewer studies were previously conducted to compare the effects of both treatment methods (mobilization and manipulation). This study specifically focuses on the comparative effects of upper thoracic and cervico-thoracic mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18-40
* Both males and Females
* Positive Hawkins and Neer's impingement test positive
* The subjects primarily report unilateral shoulder pain.

Exclusion Criteria:

* Patients with diagnosed case of co morbidities such as malignancies, RA, or fracture, that causes bilateral shoulder discomfort.
* Diagnosed case of cervical radiculopathy, glenohumeral osteoarthritis, and adhesive capsulitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  NPRS scale will be used to quantify pain intensity levels. The scale ranges from '0' for the least amount of pain "no pain" to '10' for the most extreme levels of pain "pain as severe as you can imagine". It is convenient to use NPRS for patients. Its score ranges between 0-10 (19). It is a valid and reliable tool (20).
  Reliability ranges from .67-.96 and validity ranges from 0.79-0.95
Shoulder pain and disability index SPADI | 6 weeks
  To quantify the degree to which patients affected with shoulder pain may have disability the Shoulder Pain and Disability Index (SPADI) was created. The SPADI's 13 components are split between a pain scale of five items and a disability scale of eight items. The numerical rating scale variant was created to facilitate its use and scoring (23). Reliability of SPADI is 0.92 and validity is 0.79
imagej software | 6 weeks
  It can calculate area and pixel value statistics of user-defined selections. It can measure distances and angles. It can create density histograms and line profile plots. It supports standard image processing functions such as contrast manipulation, sharpening, smoothing, edge detection and median filtering.. It has been introduced as a reliable assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Ali raza, Principal Investigator — Riphah International University; Mehreen Mazhar, Principal Investigator — Riphah inernational university
Locations (1):
- Johar pain relief center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo YP, Hsu YC, Chan KM. Epidemiology of shoulder impingement in upper arm sports events. Br J Sports Med. 1990 Sep;24(3):173-7. doi: 10.1136/bjsm.24.3.173. PMID 2078803
- [Background] Kardouni JR, Shaffer SW, Pidcoe PE, Finucane SD, Cheatham SA, Michener LA. Immediate changes in pressure pain sensitivity after thoracic spinal manipulative therapy in patients with subacromial impingement syndrome: A randomized controlled study. Man Ther. 2015 Aug;20(4):540-6. doi: 10.1016/j.math.2014.12.003. Epub 2014 Dec 22. PMID 25595413
- [Background] Michener LA, Kardouni JR, Sousa CO, Ely JM. Validation of a sham comparator for thoracic spinal manipulation in patients with shoulder pain. Man Ther. 2015 Feb;20(1):171-5. doi: 10.1016/j.math.2014.08.008. Epub 2014 Sep 6. PMID 25261090
- [Background] McCoy RC, Bittencourt E, Clifton W. Cervicothoracic Manipulation Techniques Reviewed Utilizing Three-Dimensional Spine Model. Cureus. 2019 Oct 4;11(10):e5836. doi: 10.7759/cureus.5836. PMID 31754571
- [Background] McDevitt A, Young J, Mintken P, Cleland J. Regional interdependence and manual therapy directed at the thoracic spine. J Man Manip Ther. 2015 Jul;23(3):139-46. doi: 10.1179/2042618615Y.0000000005. PMID 26309384
- [Background] Joshi S, Balthillaya G, Neelapala YVR. Immediate effects of cervicothoracic junction mobilization versus thoracic manipulation on the range of motion and pain in mechanical neck pain with cervicothoracic junction dysfunction: a pilot randomized controlled trial. Chiropr Man Therap. 2020 Aug 7;28(1):38. doi: 10.1186/s12998-020-00327-4. PMID 32762708
- [Background] Hunter DJ, Rivett DA, McKiernan S, Luton R, Snodgrass SJ. Thoracic Manual Therapy Improves Pain and Disability in Individuals With Shoulder Impingement Syndrome Compared With Placebo: A Randomized Controlled Trial With 1-Year Follow-up. Arch Phys Med Rehabil. 2022 Aug;103(8):1533-1543. doi: 10.1016/j.apmr.2022.03.003. Epub 2022 Mar 21. PMID 35331719
- [Background] Hegarty AK, Hsu M, Roy JS, Kardouni JR, Kutch JJ, Michener LA. Evidence for increased neuromuscular drive following spinal manipulation in individuals with subacromial pain syndrome. Clin Biomech (Bristol). 2021 Dec;90:105485. doi: 10.1016/j.clinbiomech.2021.105485. Epub 2021 Sep 21. PMID 34571486